CLINICAL TRIAL: NCT00442832
Title: A Phase 2, Randomized, Double Blind, Study of Intravenous TD 1792 Versus Vancomycin for Treatment of Complicated Gram Positive Skin and Skin Structure Infections
Brief Title: TD-1792 in Gram-positive Complicated Skin and Skin Structure Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0041
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Staphylococcal Skin Infection
Keywords: cSSSI; Staph; MRSA
MeSH Terms: conditions — Staphylococcal Skin Infections; Staphylococcal Infections | interventions — cefilavancin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-1792 (Experimental)
  Interventions: Drug: TD-1792
- Vancomycin (Active Comparator)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: TD-1792 — TD-1792 2 mg/kg/day IV
  Arms: TD-1792
Drug: Vancomycin — Vancomycin 1 Gm IV q 12 hrs
  Arms: Vancomycin

SUMMARY:
The purpose of this study is to determine whether TD-1792 is safe and effective when used to treat complicated skin and skin structure infections caused by Gram-positive bacteria.

DETAILED DESCRIPTION:
TD-1792 is compared to vancomycin for the treatment of cSSSI.

ELIGIBILITY:
Inclusion Criteria:

* major abscess requiring surgical incision and drainage,infected burn, deep/extensive cellulitis, infected ulcer, wound infections
* requires at least 7 days of intravenous antibiotic treatment

Exclusion Criteria:

* more than 24 hours of antibiotic therapy
* moderate or severe liver disease
* severely neutropenic
* baseline QTc > 500 msec, congenital long QT syndrome, uncompensated heart failure, uncorrected abnormal K+ or Mg++ blood levels or severe left ventricular hypertrophy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Clinical response | 7 to 14 days after last antibiotic dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Allan Churukian, National City, California, United States